CLINICAL TRIAL: NCT03301311
Title: Using Single Subject (N-of-1) Designs to Answer Patient-Identified Research Questions--Aim 1: Personalized Research on Diet in Ulcerative Colitis and Crohn's Disease
Brief Title: Personalized Research on Diet in Ulcerative Colitis and Crohn's Disease
Acronym: PRODUCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: University of California, San Francisco (Other); Seattle Children's Hospital (Other); Dayton Children's Hospital (Other); Brown University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CIN001-PRODUCE
Record Dates: First submitted 2017-09-26; First posted 2017-10-04 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Inflammatory Bowel Diseases; Crohn Disease; Ulcerative Colitis; Indeterminate Colitis
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Intervention Model Description: We are using a series of N-of-1 trials where patients alternate (cross) between the two study interventions at set intervals. N-of-1 trial results will be examined at the individual and population level (through meta-analysis of individual N-of-1 trials)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Specific Carbohydrate Diet (First) (Experimental): Participants will be following the Specific Carbohydrate Diet (SCD). Allowed foods include meat/fish/poultry, eggs, some legumes (e.g., lentils and split peas are permitted, chickpeas and soybeans are not), fully fermented yogurt, non-starchy vegetables, ripe fruit, nuts/seeds, honey and nut flours (e.g. almond flour or coconut flour). Restricted foods include all grains, milk products aside from 24-hour fermented SCD yogurt and cheeses aged greater than 30 days, starchy vegetables, processed foods with food additives and sweeteners other than honey.
  Interventions: Other: Specific Carbohydrate Diet (SCD); Other: Modified Specific Carbohydrate Diet (MSCD)
- Modified Specific Carbohydrate Diet (First) (Experimental): Participants will be following a modified Specific Carbohydrate Diet (MSCD). In addition to the foods in the SCD, allowed foods will expand to include organic rice, oats, sweet potatoes, grade A maple syrup and cocoa. Gluten, corn products, milk products (except yogurt and hard cheeses), sweeteners (except honey), and process foods are still restricted.
  Interventions: Other: Specific Carbohydrate Diet (SCD); Other: Modified Specific Carbohydrate Diet (MSCD)

INTERVENTIONS:
Other: Specific Carbohydrate Diet (SCD) — Patients will be randomized to start with either a strict SCD or modified SCD. Participants will alternate between each diet in 8-week intervals for a total duration of approximately 34 weeks. Participants will complete two 8-week intervention periods on each diet.
Other: Modified Specific Carbohydrate Diet (MSCD) — Patients will be randomized to start with either a strict SCD or modified SCD. Participants will alternate between each diet in 8-week intervals for a total duration of approximately 34 weeks. Participants will complete two 8-week intervention periods on each diet.

SUMMARY:
A series of N-of-1 trials will be used to determine the effectiveness of a specific carbohydrate diet (SCD) versus a modified SCD in patients in reducing symptoms and inflammatory burden at both the individual and population level. This is a four-year study. The study staff will recruit up to 60 patients across up to 21 sites in patients aged 7-18 with mild to moderate disease activity.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Crohn's Disease (CD) or ulcerative colitis (UC) or Indeterminate colitis (IC)
* Age 7-18 years
* Enrolled in the ImproveCareNow (ICN2) registry
* Evidence of acute inflammation and/or elevated acute phase reactant as measured by Fecal calprotectin 1.5 times the upper limit of normal, Lactoferrin 1.5 times the upper limit of normal, CRP 1.15 times the upper limit of normal, or ESR 1.15 times the upper limit of normal (based on local reference ranges) obtained within 8 weeks of enrollment.

  * Potential participants who are close to meeting one of the acute inflammation and/or elevated acute phase reactant markers and who meet all other study criteria will be considered for study participation on a case by case basis by the investigative study team in consultation with the patient's primary gastroenterologist.

Exclusion Criteria:

Complex and Unstable IBD:

* Currently or within the past 9 months has had an abscess, fistula, stricturing CD, or ostomy
* Severe disease activity as measured by a short Pediatric Crohn's Disease Activity Index (SPCDAI) score of >45 or Pediatric Ulcerative Colitis Activity Index (PUCAI) score of >60 assessed within three weeks of enrollment
* Ever had history of full colectomy
* Hospitalization or surgery planned within 3 months
* Ongoing active gastrointestinal infection
* Severe Malnutrition (BMI less than 5th percentile)
* Recent medication changes including:

  * Thiopurines, natalizumab, or methotrexate started within 8 weeks prior to enrollment
  * Anti TNF (infliximab, adalimumab) started within 8 weeks prior to enrollment
  * Vedolizumab started within 16 weeks prior to enrollment
  * Increase in corticosteroids within 4 weeks of screening or have dose >20 mg prednisone or equivalent

Evidence of Other Complicating Medical Issues:

* Other serious medical conditions, such as neurological, liver, kidney, or systemic disease
* Serious psychological or psychiatric conditions such as eating disorders or self-harm
* Pregnancy
* Tobacco, alcohol, or illicit drug abuse

Inability to Complete the Protocol

* Non-English speaking participants
* On SCD or modified SCD anytime within 8 weeks of enrollment

  * If an otherwise eligible patient is on SCD or modified SCD within 8 weeks of enrollment but they are noncompliant per the determination of the patient's dietitian/primary gastroenterologist, then this patient is eligible to participant in the study.
* Participants on a vegan diet
* Lack of smart phone and data plan for participating caregiver
* Participating in another concurrent intervention study

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 54 (Actual)
Dates: Start 2018-04-10 (Actual); Primary Completion 2020-09-08 (Actual); Study Completion 2020-09-08 (Actual)

PRIMARY OUTCOMES:
Stool frequency | Daily through study completion (34 weeks from randomization)
  Self-reported number of stools per day entered as an integer in the study mobile app
Stool Consistency | Daily through study completion (34 weeks from randomization)
  Self-reported assessment of stool consistency using the Bristol Stool Scale entered in the study mobile app
Pain Interference | Weekly through study completion (34 weeks from randomization)
  Patient reported outcome of pain interference measured using the Patient Reported Outcomes Measurement Information System (PROMIS) Pain Interference Scale on the study app. The scale includes 8 items and responses to each item are on a 0 (Never) to 4 (Almost Always) scale. Higher scores indicate greater pain interference. Look up tables provided by the PROMIS Assessment Center will be used to transform the raw score to a T-score such that 50 is the mean for the population with a standard deviation of 10.
Gastrointestinal Symptoms | Weekly through study completion (34 weeks from randomization)
  Self-reported outcome of GI symptom burden measured using the PROMIS GI Symptoms scale on the study app. The scale includes 4 items and responses to each item are on a 1 (Never) to 5 (Almost Always) scale. Higher scores indicate greater GI symptom burden. Look up tables provided by the measure developers will be used to transform the raw score to a T-score such that 50 is the mean for the population with a standard deviation of 10.
Fecal Calprotectin | At baseline and once at the end of each treatment period (weeks 10, 18, 26 and 34) for a total of 5 times
  Laboratory measurement of intestinal inflammation. Stool will be collected by participants at home and will be mailed to a central lab for processing and analysis.

SECONDARY OUTCOMES:
Provider measured disease activity | At baseline, 10 weeks and up to 2 -4 more times as standard of care visits for the duration of the study (34 weeks from randomization)
  Pediatric Ulcerative Colitis Index (PUCAI) or Short Pediatric Crohn's Index (sPCDAI) are completed by care providers at all scheduled clinic visits as part of standard of care and are entered into the ImproveCareNow (ICN) registry.
Laboratory markers of disease activity and inflammation | At baseline, 10 weeks and up to 2 -4 more times as standard of care visits for the duration of the study (34 weeks from randomization)
  C-reactive protein (CRP), erythrocyte sedimentation rate (ESR), albumin, and hematocrit as collected as part of standard of care and are entered into the ImproveCareNow (ICN) registry.
Growth | At baseline, week 4, week 10, week 12 and up to 2 -4 more times as standard of care visits for the duration of the study (34 weeks from randomization)
  Weight and height are collected at all clinic visits and at the dietitian study follow up visits (2 weeks into the first diet period of each diet). These data are entered into the ICN registry as part of regular data entry. We will calculate weight for age Z-scores for all entries during study period. The age-specific mean and standard deviation from U.S. population norms will be used to calculate Z-scores using the Centers for Disease Control Epi-Info program.
Short Crohn's Disease Activity Index (sCDAI) | Weekly through study completion (34 weeks from randomization)
  The short Crohn's disease activity index (sCDAI) will be used to assess disease activity based on self-report via the study app. For the sCDAI, items assess general well-being, abdominal pain, and liquid stools. Respondents are asked to report on symptoms for the previous 24 hour period. Scores are calculated based on a published algorithm.
Pediatric Ulcerative Colitis Activity Index (PUCAI) | Weekly through study completion (34 weeks from randomization)
  A self-reported version of the Pediatric Ulcerative Colitis Activity Index (PUCAI) will be used to assess disease activity based on self-report via the study app. For the PUCAI, respondents are asked to report on abdominal pain, bloody stools, stool consistency, stool frequency, nocturnal stools, and activity level over the prior 24-hours. A weighted, summed score is calculated with higher scores indicating worse disease (score range 0-85).

CONTACTS AND LOCATIONS:
Overall Officials: Heather C Kaplan, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Lisa Opipari-Arrigan, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (20):
- United States (20):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Children's Hospital of Los Angeles, Los Angeles, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Lucile Packard Children's Hospital, Palo Alto, California
  - University of California San Francisco Benioff Children's Hospita;, San Francisco, California
  - Nemours, Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Nemours Children's Speciality Care, Jacksonville, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - GI Care for Kids, Atlanta, Georgia
  - Riley Hospital for Children, Indianapolis, Indiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Children's Mercy Hospital, Kansas City, Missouri
  - Levine Children's Hospital, Charlotte, North Carolina
  - Nationwide Children's Hospital, Columbus, Ohio
  - Oregon Health Sciences University, Portland, Oregon
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - UT Soutwestern Medical Center, Dallas, Texas
  - Pediatric Specialists of Virginia, Fairfax, Virginia
  - Children's Hospital of the King's Daughters, Norfolk, Virginia
  - Seattle Children's, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
We intend to provide access to the de-identified, HIPAA-compliant databases as required within a year after the study has been completed. Data plans, analysis plans, data dictionaries, study manuals and annotated case report forms will be made available, upon request, in a read-only format (PDF). Each dataset will be accompanied by appropriate documentation listing each variable, variable definition, decode values (if appropriate), an indication of the variable as a source collected or derived variable, and derivation algorithms for any derived values.
  Datasets will be available as SAS, SAS transport, XML or CSV with labels. Other formats may be created if requested. All necessary security measures will be taken to ensure patient privacy and confidentiality, and details on how data may be used, including the use of de-identified data sets, will be included in the informed consent.
Supporting Information: SAP
Time Frame: Within a year after study completion.

REFERENCES:
- [Result] Kaplan HC, Opipari-Arrigan L, Yang J, Schmid CH, Schuler CL, Saeed SA, Braly KL, Chang F, Murphy L, Dodds CM, Nuding M, Liu H, Pilley S, Stone J, Woodward G, Yokois N, Goyal A, Lee D, Yeh AM, Lee P, Gold BD, Molle-Rios Z, Zwiener RJ, Ali S, Chavannes M, Linville T, Patel A, Ayers T, Bassett M, Boyle B, Palomo P, Verstraete S, Dorsey J, Kaplan JL, Steiner SJ, Nguyen K, Burgis J, Suskind DL; ImproveCareNow Pediatric IBD Learning Health System. Personalized Research on Diet in Ulcerative Colitis and Crohn's Disease: A Series of N-of-1 Diet Trials. Am J Gastroenterol. 2022 Jun 1;117(6):902-917. doi: 10.14309/ajg.0000000000001800. Epub 2022 Apr 20. PMID 35442220

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-31): https://cdn.clinicaltrials.gov/large-docs/11/NCT03301311/Prot_SAP_006.pdf